CLINICAL TRIAL: NCT03942900
Title: Immunomonitoring and Biomarker Research Based on Tumor and Blood Samples in Patients With Squamous Cell Anal Carcinoma
Brief Title: Immunomonitoring and Biomarker Research in Patients With Squamous Cell Anal Carcinoma
Acronym: LAND
Status: Withdrawn | Type: Observational
Why Stopped: Study not submitted to regulatory authorities
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2018/381
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Anal Canal Cancer
Keywords: locally advanced SCCA; DCF; radiotherapy; nivolumab; biomarkers
MeSH Terms: conditions — Anal Canal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A tumor biopsy or archived tumor sample will be mandatory at baseline. Tumor samples will be collected for HPV, p53 testing and translational research.
  * Biomonitoring blood sample will be collected: 6 EDTA (ethylenediaminetetraacetic acid) tubes (6 mL) for PBMC, 1 EDTA tube (6 mL) for plasma freezing and 2 EDTA tubes (4 mL) for circulating tumor DNA (ctDNA):
    * at baseline,
    * at first tumor assessment (phase 2 in OPTIMANAL study),
    * at second tumor assessment (phase 4 in OPTIMANAL study),
    * at end-point visit
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort LAND: Patients enrolled in OPTIMANAL clinical trial
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — * Biomonitoring blood sample will be collected: 6 EDTA tubes (6 mL) for PBMC (peripheral blood mononucleated cell), 1 EDTA tube (6 mL) for plasma freezing and 2 EDTA tubes (4 mL) for ctDNA:
    * at baseline,
    * at first tumor assessment (phase 2 in OPTIMANAL study),
    * at second tumor assessment (phase 4 in OPTIMANAL study),
    * at end-point visit.
  * A tumor biopsy or archived tumor sample will be mandatory at baseline.

SUMMARY:
Even if squamous cell carcinoma of the anal canal (SCCA) is a rare disease, its incidence increases worldwide. SCCA is mostly induced by Human papillomavirus (HPV) infections and HPV-related oncoproteins (E6 and E7) are expressed in more than 90% of SCCA. T stage and N stage are recognized prognostic factors for local and/or distant recurrence in SCCA patients treated by chemoradiotherapy. In fact, ≥T3 or ≥N1 anal cancers are associated with as high as 50% of disease recurrence rate at 2 years.

The University Hospital of Besançon with the Gercor conducted a prospective clinical trial (Epitopes HPV02 study) including 69 advanced SCCA patients and established a new standard of care based on Docetaxel, Cisplatin and 5-FU (5-FluoroUracil) chemotherapy (DCF). Among 69 patients treated with DCF regimen, 66 patients were evaluable for efficacy end-points. The objective response rate was 86% including 44% of complete response, and 47% of patients were progression-free at 12 months of follow-up from the first cycle of DCF treatment. Thus, the "Epitopes-HPV02" trial has demonstrated a high response rate of the DCF regimen with a higher than expected 12 months progression-free survival rate.These results raised the hypothesis of DCF being an immunogenic chemotherapy and in that demonstrating a possibly new role of taxane-based chemotherapy in SCCA patients. More than 50% of patients in complete remission had a detectable immunological response against peptides derived from HPV oncoproteins (E6 or E7) or from the telomerase antigen (which is transactivated by E6).

LAND study will enroll patients with locally advanced SCCA enrolled in OPTIMANAL clinical trial. OPTIMANAL study will assess the feasibility and efficacy to combine nivolumab to mDCF chemotherapy, followed by the standard chemo-radiotherapy, in high risk locally advanced SCCA patients with T3/T4 N1a or N1b/N1c disease.

LAND study is an exploratory translational study, which will analyze the biological mechanisms of action and our ability to track the immune responses against HPV and telomerase. The investigator group will take advantage of the presence of HPV antigens in most patients to set up a specific immunomonitoring program based on tumor samples and blood-derived lymphocytes to better understand the potential synergisms between immunogenic chemotherapy and anti-PD1 (Programmed Death-1), and to identify valuable biomarkers of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years,
2. Patients enrolled in OPTIMANAL trial
3. Signed and dated informed consent for LAND-translational study
4. Histologically proved squamous cell anal carcinoma.

Exclusion Criteria:

1. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study,
2. Patient under guardianship, curators or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced squamous cell anal carcinoma enrolled in OPTIMANAL clinical trial, and given consent for LAND-translational study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Peripheral CD4 anti-telomerase immunity and MDSC (Myeloid-Derived Suppressor Cells) analysis | 24 months
  Correlation of both peripheral CD4 anti-telomerase immunity and MDSC with progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BORG, Pr, Study Director — CHU Besançon
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim S, Jary M, Andre T, Vendrely V, Buecher B, Francois E, Bidard FC, Dumont S, Samalin E, Peiffert D, Pernot S, Baba-Hamed N, El Hajbi F, Bouche O, Desrame J, Parzy A, Zoubir M, Louvet C, Bachet JB, Nguyen T, Abdelghani MB, Smith D, De La Fouchardiere C, Aparicio T, Bennouna J, Gornet JM, Jacquin M, Bonnetain F, Borg C. Docetaxel, Cisplatin, and 5-fluorouracil (DCF) chemotherapy in the treatment of metastatic or unresectable locally recurrent anal squamous cell carcinoma: a phase II study of French interdisciplinary GERCOR and FFCD groups (Epitopes-HPV02 study). BMC Cancer. 2017 Aug 25;17(1):574. doi: 10.1186/s12885-017-3566-0. PMID 28841909
- [Background] Bernard-Tessier A, Jeannot E, Guenat D, Debernardi A, Michel M, Proudhon C, Vincent-Salomon A, Bieche I, Pierga JY, Buecher B, Meurisse A, Francois E, Cohen R, Jary M, Vendrely V, Samalin E, El Hajbi F, Baba-Hamed N, Borg C, Bidard FC, Kim S. Clinical Validity of HPV Circulating Tumor DNA in Advanced Anal Carcinoma: An Ancillary Study to the Epitopes-HPV02 Trial. Clin Cancer Res. 2019 Apr 1;25(7):2109-2115. doi: 10.1158/1078-0432.CCR-18-2984. Epub 2018 Nov 30. PMID 30504426
- [Result] Kim S, Francois E, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, De La Fouchardiere C, Smith D, Deberne M, Spehner L, Badet N, Adotevi O, Anota A, Meurisse A, Vernerey D, Taieb J, Vendrely V, Buecher B, Borg C. Docetaxel, cisplatin, and fluorouracil chemotherapy for metastatic or unresectable locally recurrent anal squamous cell carcinoma (Epitopes-HPV02): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2018 Aug;19(8):1094-1106. doi: 10.1016/S1470-2045(18)30321-8. Epub 2018 Jul 2. PMID 30042063